CLINICAL TRIAL: NCT01394627
Title: Hypoglycemia and the Mineralocorticoid Receptor
Acronym: HypoMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Robert Wood Johnson Foundation (Other); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Gail Kurr Adler, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2010P002054; K24HL103845 (NIH); R01HL109634 (NIH); T32HL007609 (NIH)
Record Dates: First submitted 2011-07-11; First posted 2011-07-14 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eplerenone (Experimental): hypoglycemia (50 mg/dl) with pretreatment with two doses of eplerenone (100 mg of eplerenone per dose)
  Interventions: Drug: Eplerenone
- placebo (Placebo Comparator): hypoglycemia of 50 mg/dl plus placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eplerenone — 100mg x 2
  Arms: Eplerenone
Drug: Placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to look at whether blockade of the mineralocorticoid receptor will result in changes in the cardiovascular and inflammatory response to hypoglycemia.

DETAILED DESCRIPTION:
The effect of ongoing hypoglycemia on cardiovascular autonomic function is unclear and the focus of this protocol. In our preliminary studies, the investigators demonstrated that baroreflex sensitivity is impaired during hypoglycemia in healthy individuals. Treatment with eplerenone (200mg total administered in two doses in the 15 hours prior to the hypoglycemic clamp) prevented this impairment.

The study is based on the overarching hypothesis that hypoglycemia leads to increases in aldosterone/mineralocorticoid receptor (MR) activity and increased cardiovascular injury.

This study will address the following Specific Aims:

To test the hypothesis that MR blockade will reduce the adverse effects of hypoglycemia on inflammation and on autonomic control of cardiovascular function.

The investigators will determine the effects of hypoglycemia (50 mg/dl for 2.0 hours) on the blood inflammatory factor interleukin-6 levels, and on cardiovascular autonomic function (baroreflex sensitivity) in each subject under two conditions - pretreatment with MR blockade (eplerenone) and pretreatment with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Males and females age 18 to 40 years

Exclusion Criteria:

* Pregnancy
* Lactation
* Menopause
* Any medical condition other than treated hypothyroidism.
* Alcoholism
* Active tobacco use
* In all subjects, any individuals on oral, injected, inhaled or topical corticosteroids within the last year or oral contraceptives within the past 3 months will be excluded.
* Use of medications other than physiological thyroxine replacement
* Serum potassium >5.0 mmol/L
* Estimated glomerular filtration rate < 60 mL/min

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail K Adler, MD, Principal Investigator — Brigham and Women's Hospital; Gail K Adler, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Rao AD, Bonyhay I, Dankwa J, Baimas-George M, Kneen L, Ballatori S, Freeman R, Adler GK. Baroreflex Sensitivity Impairment During Hypoglycemia: Implications for Cardiovascular Control. Diabetes. 2016 Jan;65(1):209-15. doi: 10.2337/db15-0871. Epub 2015 Oct 5. PMID 26438610

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Period 1) /Washout (Period 2)/Eplerenone (Period 3): hypoglycemia of 50 mg/dl with 1 day of placebo pretreatment
  then after 1-3 month washout
  hypoglycemia of 50 mg/dl with 1 day of eplerenone (100 mg x 2) pretreatment
- Eplerenone (Period 1) /Washout (Period 2)/Placebo (Period 3): hypoglycemia of 50 mg/dl with 1 day of eplerenone (100 mg x 2) pretreatment
  then after 1-3 month washout
  hypoglycemia of 50 mg/dl with 1 day of placebo pretreatment
Period: First Intervention (1 Day)
Arm/Group | Placebo (Period 1) /Washout (Period 2)/Eplerenone (Period 3) | Eplerenone (Period 1) /Washout (Period 2)/Placebo (Period 3)
Started | 8 | 13
Completed | 8 | 12
Not Completed | 0 | 1
Not completed — poor intravenous access | 0 | 1
Period: Washout (1-3 Months)
Arm/Group | Placebo (Period 1) /Washout (Period 2)/Eplerenone (Period 3) | Eplerenone (Period 1) /Washout (Period 2)/Placebo (Period 3)
Started | 8 | 12
Completed | 7 | 12
Not Completed | 1 | 0
Not completed — concurrent enrollment in another study | 1 | 0
Period: Second Intervention (1 Day)
Arm/Group | Placebo (Period 1) /Washout (Period 2)/Eplerenone (Period 3) | Eplerenone (Period 1) /Washout (Period 2)/Placebo (Period 3)
Started | 7 | 12
Completed | 7 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 12
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cardiovascular Autonomic Function
Description: Modified oxford procedures was performed in duplicate immediately prior to start of the hypoglycemic clamp and during the last 30 min of the clamp (i.e. during the last 30 min of exposure to 2 hours of hypoglycemia).. We calculated the baroreflex sensitivity (the relationship between RR interval and change in systolic blood pressure defined as the change in the inter-beat cardiac interval in milliseconds per unit change in blood pressure in mmHg) at each time point and then the change in baroreflex sensitivity (BRS during hypoglycemia minus BRS at baseline)
Time Frame: Baseline and 2 hours after hypoglycemia
Population: We included the 13 subjects who completed each arm, had usable baroreflex sensitivity data for both treatments (placebo and eplerenone), and achieved a blood sugar during hypoglycemia of less than or equal to 3.0 mmol/L for each clamp.
Measure: Mean (Standard Deviation); unit: ms/mmHg
Groups:
- Placebo: hypoglycemia of 50 mg/dl plus placebo
  Placebo
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 13 | 13
ms/mmHg | -16.00 (18.39) | -16.59 (16.77)

2. Secondary Outcome: Change From Baseline in Inflammation
Description: Change in interleukin-6
Time Frame: Baseline and 2 hours after hypoglycemia
Population: We included the 17 subjects who completed each arm and had interleukin-6 data for both arms (placebo and eplerenone). We calculated the change in IL-6 as IL-6 during hypoglycemia minus IL-6 at baseline.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 17 | 17
pg/ml | 2.03 (1.27) | 2.61 (2.63)

ADVERSE EVENTS:
Groups:
- Eplerenone: hypoglycemia (50 mg/dl) with pretreatment with two doses of eplerenone (100 mg of eplerenone per dose) Eplerenone: 100mg x 2
Arm/Group | Eplerenone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes